CLINICAL TRIAL: NCT04463862
Title: Air Pollution and COVID-19 Mortality in Geriatric Patients: a Multicenter Study
Brief Title: COVID - AirPollution
Status: Completed | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 7922
Record Dates: First submitted 2020-07-08; First posted 2020-07-09 (Actual); Last update posted 2021-06-25 (Actual); Status verified 2021-06

CONDITIONS: COVID-19 Confirmed Cases; COVID-19 Mortality
Keywords: Air pollution; COVID-19; Respiratory viral diseases; PM- NO2-Ozone
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epidemiological data have related particulate matter (PM), nitrogen dioxide (NO2) and ozone (O3) to COVID-19 morbidity and mortality at the population level. Air pollution may be related to an increase in the COVID-19 severity and lethality through its impact on chronic diseases such as cardiovascular and respiratory diseases and diabetes that are also the main comorbidities associated with COVID-19. Epidemiological studies using individual data are needed to provide more precise estimate of the association between air pollution exposure and COVID-19. In this multicenter prospective study, the investigators will analyze the number of deaths in COVID-19 confirmed cases in geriatric patients according to long-term exposure to air pollution, taking into account confounders such as diabetes, hypertension, age, and BMI. Exposure to air pollution will be estimated as the mean concentration of air pollutants at the residential address during the previous two years. In addition, the investigators will explore the relationship between short-term variations in air pollutants, relative humidity, temperature, UV radiations, pollen and the occurrence of COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 60 years old (or dementia patient over 50 years old)
* Patient hospitalized in a geriatric department over the period from 2020/01/01 to 2020/06/01
* Patient who underwent RT-PCR SARS-CoV-2
* Patient (or trusted person/ legal guardian/curator, if applicable) who has given consent to the re-use of his/her data (patient data) for research purposes

Exclusion Criteria:

None

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted in geriatric departments between 2020/01/01 to 2020/06/01
Sampling Method: Non-Probability Sample
Enrollment: 660 (Actual)
Dates: Start 2020-06-04 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

PRIMARY OUTCOMES:
COVID-19 related-mortality | COVID-19 mortality between 2020/01/01 and 2020/06/01
  Association between COVID-19 related-mortality and air pollutants concentrations estimated at the residential address of geriatric patients during the last 2 years ( from 2018/01/01 to 2019/12/31)

SECONDARY OUTCOMES:
COVID-19 confirmed cases | COVID-19 confirmed cases between 2020/01/01 and 2020/06/01
  Association between short- term variations in air pollutants, temperature, humidity, UV, pollens and the occurrence of COVID-19 confirmed cases.
  Short-term variations are defined as changes in air pollutants concentrations, temperature, humidity and pollen during the 20 days preceding the hospitalization.

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric BLANC, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (8):
- Unité de neurologie-gériatrie, Hôpital Erasme, Cliniques Universitaires de Bruxelles, Brussels, Belgium
- France (7):
  - Unité de soins palliatifs gériatriques, Centre Hospitalier Départemental de Bischwiller, Bischwiller
  - Service de Gériatrie, Centre Hospitalier Départemental de Vendée, La Roche-sur-Yon
  - Service de médecine aigüe gériatrique, Hôpital Nord Laennec, Hôpitaux Universitaires de Nantes, Nantes
  - Service de Gériatrie, Hôpitaux Bichat et Bretonnaux, Assistance Publique des Hôpitaux de Paris, Paris
  - Service de Médecine Interne et Gériatrie, Hôpitaux Universitaires de Reims, Reims
  - Service de Gériatrie, Hôpital de la Robertsau, Hôpitaux Universitaires de Strasbourg, Strasbourg
  - Service de médecine gériatrique, Hôpitaux Universitaires de Tours, Tours

IPD SHARING:
Plan to Share IPD: No